CLINICAL TRIAL: NCT02188537
Title: Nelfinavir as Bortezomib-sensitizing Drug in Patients With Proteasome Inhibitor-nonresponsive Myeloma. A Multicenter Phase II Trial
Brief Title: Nelfinavir as Bortezomib-sensitizing Drug in Patients With Proteasome Inhibitor-nonresponsive Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 39/13 - FORTUNE; SNCTP000001061 (Registry Identifier: SNCTP)
Record Dates: First submitted 2014-07-03; First posted 2014-07-11 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Myeloma
Keywords: Myeloma; proteasome inhibitor-nonresponsive myeloma; Nelfinavir; bortezomib; bortezomib-sensitizing drug
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Nelfinavir; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir, Bortezomib, Dexamethasone (Experimental): The trial is designed as an "add-on" therapy, where nelfinavir is added to the approved bortezomib-containing therapy. Bortezomib and dexamethasone background treatment will be given in the Swissmedic-approved dose and schedule and according to international therapeutic standard.
  Interventions: Drug: Nelfinavir; Drug: bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Nelfinavir — Nelfinavir 2x 2500 mg p.o. days 1 - 14
  Other Names: Viracept
Drug: bortezomib — Bortezomib 1.3 mg/m2 i.v. or s.c. days 1, 4, 8, 11
  Other Names: Velcade®
Drug: Dexamethasone — Dexamethasone 20 mg p.o. days 1-2, 4-5, 8-9, 11-12

SUMMARY:
Trial objectives:

To decide whether the addition of nelfinavir to the approved antimyeloma therapy with bortezomib and dexamethasone has sufficient activity in proteasome inhibitor-resistant myeloma patients to merit further clinical investigation in a prospective controlled trial.

Additional research questions:

To collect myeloma cell samples from proteasome inhibitor-resistant myeloma patients for the assessment of the biology of proteasome inhibitor resistance and the identification of predictive markers for response to nelfinavir-based antimyeloma therapy.

DETAILED DESCRIPTION:
Trial objectives:

To decide whether the addition of nelfinavir to the approved antimyeloma therapy with bortezomib and dexamethasone has sufficient activity in proteasome inhibitor-resistant myeloma patients to merit further clinical investigation in a prospective controlled trial.

Additional research questions:

To collect myeloma cell samples from proteasome inhibitor-resistant myeloma patients for the assessment of the biology of proteasome inhibitor resistance and the identification of predictive markers for response to nelfinavir-based antimyeloma therapy.

Primary endpoint:

Response rate based on best response observed during the trial

Selection of patients:

* Patients with multiple myeloma based on standard IMWG criteria, who have received at least one prior line of chemotherapy
* Previously exposed to or intolerant to at least one immunomodulatory drug (IMID) (thalidomide, lenalidomide, pomalidomide)
* Refractory to their most recent proteasome inhibitor-containing regimen or progressed during or within 60 days after proteasome inhibitor-containing therapy
* A bortezomib-based therapy in agreement with Swissmedic approval is indicated and intended
* Measurable disease based on serum paraprotein or free light chain levels
* Adequate hematological, hepatic and renal functions
* Absence of myeloma within the CNS
* No significant neuropathy
* No concomitant use of listed drugs which cannot be replaced or paused during trial treatment (Amiodarone, Pimozide, quinidine and its derivatives, ergot derivatives (dihydroergotamine, ergotamine, ergonovine, methylergonovine), triazolam, midazolam, sildenafil, alfuzosin)

Trial Schedule and Duration:

The inclusion of patients is planned to start in Q3 2014 and will stop after the inclusion of 34 evaluable patients, which is expected in Q1 2016. End of trial treatment is expected for Q3 2016. Trial termination (last patient last visit) is expected to be in 2017.

Accrual may be interrupted or the trial may be stopped early based on the results of an interim analysis or if new scientific data become available which change assessment of risk/benefit.

Trial product:

For this trial nelfinavir is the IMP. Bortezomib (Velcade®) and dexamethasone are not investigational drugs in the context of this trial, but will be administered as a background medication.

Trial Treatment:

The trial treatment is designed as an "add-on" therapy, where nelfinavir is added to the approved bortezomib therapy. Bortezomib and dexamethasone background treatment will be given in the approved dose and schedule (either i.v. or s.c), as per Swissmedic label and international therapeutic standard, in combination with 2500 mg Nelfinavir bid p.o. day 1-14 for 6 cycles of 21 days.

Measurements and procedures:

Before the trial treatment Clinical examination; blood analyses; imaging investigations if applicable (e.g. bone X-ray or computer tomography, MRI); electrocardiogram; evaluation of the quality of life with a patient's questionnaire; pregnancy test for women in child-bearing age; optional: a bone marrow sample is taken for translational research. Aside from the electrocardiogram, the pregnancy test and the quality of life questionnaire, all the pre-treatment assessments performed within the frame of the trial are also routinely performed for the medical care of patients with multiple myeloma outside of a trial.

During the trial treatment Clinical examination and blood analyses for the control of safety laboratory parameters; evaluation of the quality of life with a patient's questionnaire will be performed after completion of 3 cycles of therapy. Besides the quality of life questionnaire, all assessments would also be performed routinely outside of the trial.

After the trial treatment Clinical examination and blood analyses for the control of safety laboratory parameters; these investigations will be performed within 1 month after treatment end, premature interruption or before the administration of a new antimyeloma therapy. These assessments are routinely done also outside of the trial.

Statistical Considerations:

The Simon's two-stage design will be used. A response rate of 15% or less is considered uninteresting and 35% or higher is promising. The trial will be stopped early if the treatment appears unpromising at the end of the first stage. To allow patient accrual while waiting for the stage-1 results, the design is modified according to Herndon's approach.

With a significance level of 5% and a power of 80%, a total of 34 patients are required with 10 patients in the first stage and 24 patients in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* Patient must give written informed consent prior to any protocol-specific procedure.
* Patient was diagnosed with multiple myeloma based on standard IMWG criteria, and has received at least one previous line of chemotherapy.
* Patient has been exposed to or is intolerant to at least one IMID (thalidomide, lenalidomide, pomalidomide).
* A therapy with bortezomib in the approved dose and schedule, based on Swissmedic approval (treatment of patients with relapsed/refractory multiple myeloma who have received at least one prior line of therapy), is indicated and intended.
* Patient is refractory to his/her most recent proteasome inhibitor-containing regimen, based on divers criteria.
* WHO performance status ≤ 3.
* Age ≥ 18 years.
* Adequate hematological values: platelets ≥ 50 x 109/L, hemoglobin ≥ 80 g/L (both may be achieved by transfusion).
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN (for patients with suspected hemolysis: direct bilirubin ≤ 1.5 x ULN), ALT ≤ 3 x ULN (≤ 5 x ULN if liver infiltration by myeloma suspected, based on imaging results).
* Calculated creatinine clearance ≥ 15 mL/min, according to the formula of Cockcroft-Gault, see Appendix 1).
* Women are not breastfeeding. Women with child-bearing potential are using effective contraception (see 9.8), are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. A negative pregnancy test before inclusion (within 7 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and during 12 months thereafter.
* Completed baseline QoL questionnaire.

Exclusion Criteria:

* Evidence of ongoing uncontrolled systemic infections.
* History of chronic active HCV or HBV.
* Evidence of myeloma within the CNS.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out quality of life (QoL) forms, or interfering with compliance for oral drug intake.
* Exposure to another experimental drug within 3 weeks prior to trial entry.
* Any serious underlying medical condition (at the judgment of the investigator) which may impair the ability of the patient to participate in the trial, in particular any uncontrolled clinically significant active disease (e.g. active autoimmune disease, uncontrolled diabetes, uncontrolled cardiac disease).
* Non-hematologic active malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
* Concomitant use of other anti-cancer medication or radiotherapy except for local pain control. The use of bisphosphonates is allowed.
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to enrollment.
* Known hypersensitivity to bortezomib or nelfinavir or hypersensitivity to components of these drugs.
* Any psychological, familial, sociological or geographical condition likely hampering compliance with the trial protocol and follow-up.
* Patient who takes the following drugs during the trial therapy, which cannot be replaced or paused.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Response rate based on best response observed during the trial | end of cycle 6 (at week 19)

SECONDARY OUTCOMES:
Adverse events | end of cycle 6 (at week 19)
Proportion of patients achieving at least a minor response | end of cycle 6 (at week 19)
Disease control rate (no evidence of disease progression for at least 3 cycles) | end of cycle 6 (at week 19)
Time from registration to the start of the next new antimyeloma therapy or death from any cause | end of cycle 6 (at week 19)
Progressive disease under trial treatment | end of cycle 6 (at week 19)
Quality of life | day 1 of cycle 4 (week 10)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Driessen, Prof MD, Study Chair — Cantonal Hospital of St. Gallen; Panagiotis Samaras, MD, Study Chair — Universitätsspital Zürich
Locations (12):
- Switzerland (12):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico Svizzera Italiana IOSI, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Driessen C, Muller R, Novak U, Cantoni N, Betticher D, Mach N, Rufer A, Mey U, Samaras P, Ribi K, Besse L, Besse A, Berset C, Rondeau S, Hawle H, Hitz F, Pabst T, Zander T. Promising activity of nelfinavir-bortezomib-dexamethasone in proteasome inhibitor-refractory multiple myeloma. Blood. 2018 Nov 8;132(19):2097-2100. doi: 10.1182/blood-2018-05-851170. Epub 2018 Sep 20. No abstract available. PMID 30237154